CLINICAL TRIAL: NCT02103842
Title: Omega-3 Fatty Acids to Combat Sarcopenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ian R. Lanza, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-000639
Record Dates: First submitted 2014-03-18; First posted 2014-04-04 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omega-3 fatty acids (Experimental): Participants will take 3.9g/day of Eicosapentaenoic acid and docosahexaenoic acid for 4 months
  Interventions: Drug: Omega-3 fatty acids

INTERVENTIONS:
Drug: Omega-3 fatty acids

SUMMARY:
The purpose of this study is to determine how omega-3 fatty acids influence muscle protein metabolism and mitochondrial physiology in the context of human aging.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 or 65-85 years

Exclusion Criteria:

1. Current use of omega-3 nutritional supplements
2. Fasting plasma glucose ≥126 mg/dL
3. Active coronary artery disease
4. Participation in structured exercise (>3 times per week for 30 minutes or longer)
5. Smoking
6. Medications known to affect muscle metabolism (e.g., beta blockers, corticosteroids, tricyclic-antidepressants, benzodiazepines, opiates, barbiturates, anticoagulants)
7. Renal failure (serum creatinine > 1.5mg/dl)
8. Chronic active liver disease (Bilirubin > 17mmol/L, AST>144IU/L, or ALT>165IU/L)
9. Anti-coagulant therapy (warfarin/heparin)
10. INR >3
11. Use of systemic glucocorticoids
12. Chronic use of NSAIDS or aspirin
13. Pregnancy or breastfeeding
14. Alcohol consumption greater than 2 glasses/day
15. Hypothyroidism
16. Fish or shellfish allergy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Muscle protein synthesis | Baseline and following 4 months intervention
  Skeletal muscle protein synthesis will be measured from the rate of incorporation of infused amino acids measured by mass spectrometry.
Change in Muscle mitochondrial function | Baseline and following 4 months intervention
  Mitochondrial function will be measured in isolated mitochondria by high-resolution respirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Lanza, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States